CLINICAL TRIAL: NCT05077579
Title: Neuroinflammation and Alzheimer's Disease Imaging Biomarkers in Midlife Obesity
Brief Title: Alzheimer"s Imaging Biomarkers in Obesity
Status: Recruiting | Type: Observational
Sponsor: Cyrus A Raji (Other)
Responsible Party: Sponsor-Investigator, Cyrus A Raji, Assoc. Prof of Radiology, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Other Study IDs: 202102186
Record Dates: First submitted 2021-06-25; First posted 2021-10-14 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Disease; Obesity; Metabolic Disease
MeSH Terms: conditions — Alzheimer Disease; Obesity; Metabolic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- metabolically abnormal overweight & obese
- metabolically normal overweight
- obese and metabolically normal lean

SUMMARY:
High body fat at midlife, as evidenced by overweight or obese body mass index (BMI), is increasingly understood as a risk factor for Alzheimer's disease. However, the underlying processes and mechanisms that may underlie this risk remains unknown. With this project, the Investigator proposes to create a new cohort of cognitively normal 120 midlife individuals, age 40-60 years. The investigator and research staff will characterize the participant's overweight or obese status using metabolic tests including, an oral glucose tolerance test, fasting plasma insulin, fasting plasma glucose, and hemoglobin A1c measurements. This testing will generate categories of metabolically abnormal overweight and obese (MAOO), metabolically normal overweight and obese (MNOO), and metabolically normal lean participants (MNLP). Research staff will evaluate differences between these groups on neuroimaging with the newer classification framework of Alzheimer's biomarkers with amyloid (A), tau (T), and neurodegeneration (N), or ATN. Neurodegeneration will be assessed by atrophy on brain MRI as reflected by regional volumes on Freesurfer. Staff will also evaluate MR neuroimaging markers for neuroinflammation using a newer method called diffusion basis spectrum imaging (DBSI), developed at the Mallinckrodt Institute of Radiology at Washington University in St. Louis in collaboration with The Charles F. and Joanne Knight Alzheimer's Disease Research Center (Knight ADRC).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female, 40-60 years of age and any race;
2. MMSE = or greater than 25 or a Clinical Dementia Rating Scale (CDR)=0;
3. Willing and able to undergo MRI
4. Willing to complete PET scans, including [11C]PiB and 18F-AV-1451 (Flortaucipir) radioactive tracer injection under protocols IRB #201409014 & 201906028
5. Willing to participate in the metabolic subtyping of metabolically normal or abnormal overweight or obese status for the following three groups:

   a. Group 1: MAOO criteria: i. BMI ≥25 but <45 kg/m2; ii. Maximum body circumference < 165 cm to ensure participants fit into the PET/CT and MR scanners; iii. Fasting blood glucose: ≥100 mg/dl or blood glucose 2 h after an OGTT: ≥140 or fasting insulin: >20 µu/ml;

   b. Group 2: MNOO criteria: i. BMI ≥ 25 but <45 kg/m2; ii. Maximum body circumference < 165 cm to ensure participants fit into the PET/CT and MR scanners; iii. Blood glucose 2 h after an OGTT: iv. HbA1c < 5.7% v. Fasting insulin: < 20 µu/ml;

   c. Group 3: MNLP criteria: i. BMI ≥18.5 but < 25.0 kg/m2; ii. Maximum body circumference < 165 cm to ensure subjects fit into the PET/CT and MR scanners; iii. Fasting blood glucose: < 100 mg/dl; iv. Blood glucose 2 h after an OGTT: < 140 mg/dl; v. HbA1c < 5.7% vi. Fasting insulin: < 20 µu/ml;

Exclusion Criteria:

1. Any condition that in the opinion of the Investigator or designee could increase the risk to the participant, limit the participant's ability to tolerate the research procedures or interfere with the collection of the data, (e.g., currently taking a drug for treatment of obesity);
2. Intend to have bariatric surgery;
3. Inability to tolerate to lie still during the scanning procedures (e.g., severe, chronic back pain);
4. Severe claustrophobia;
5. Women who are currently pregnant or breast-feeding;
6. Currently receiving an active obesity study drug (or placebo) or in an obesity clinical trial;
7. Laboratory Evaluations exclusion: • Oral glucose tolerance test should not be performed in patients who already fulfill the criteria for diabetes mellitus. These include: - History of Type 1 or 2 diabetes mellitus - Prior documentation of a fasting plasma glucose >7.0 mmol/L or two or more occasions or clinical symptoms of diabetes e.g. polydipsia, polyuria, ketonuria and rapid weight loss with a random plasma glucose of >11.1 mmol/L • Other contraindications for venous access as part of OGTT or blood draws: - Venous fibrosis or shunt grafts in both upper extremities - Ongoing cellulitis or infection, particularly in the upper extremities. - Presence of a hematoma at the site of vascular access. - History of hypoglycemic encephalopathy that can occur with prolonged fasting
8. MRI exclusion: • Contraindications to MRI (e.g., certain incompatible electronic medical devices that make it potentially unsafe for the individual to participate). All participants must be willing to undergo at least two MRI screenings, supervised by Level II MRI personnel as designated by the American College of Radiology (ACR).

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We currently have IRB-approved protocols covering ongoing imaging that meet the eligibility criteria. The Washington University Knight Alzheimer's Disease Research Center and the Center for Human Nutrition will refer participants . The Knight ADRC primarily recruits participants by means of word of mouth and public service announcements from the greater metropolitan St. Louis area. We will also coordinate these efforts with the Center for Human Nutrition to maximize potential participants from their studies. A small percentage (~17%) of participants are referred by Washington University physicians. The Research Participant Registry/Volunteer for Health (VFH) Program at Washington University in St. Louis (https://vfh.wustl.edu) will also be utilized.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Aim - increased atrophy in MAOO compared to MNOO and MNLP participants | 10 hours
  we hypothesize increased atrophy in MAOO compared to MNOO and MNLP particularly in regions important for AD pathology such as the hippocampus and hippocampal sub-regions. These will be measured through the results of the blood tests, MRI scan & data from the PET scans.

SECONDARY OUTCOMES:
Aim 2- higher burden of white matter neuroinflammation on DBSI | 10 hours
  We hypothesize a higher burden of white matter neuroinflammation on DBSI in MAOO in relation to other overweight and obese groups. The MRI scan will be used to measure these outcomes.
Aim 3-increased amyloid and tau deposition on brain | 10 hours
  We hypothesize increased amyloid and tau deposition on brain PET in MAOO versus other groups. The PET scan data will be used to measure these outcomes.

OTHER OUTCOMES:
Sub-aims-sex differences in atrophy and neuroinflammation | 10 hours
  Will examine sex differences in atrophy and neuroinflammation. We will also investigate sex differences in amyloid and tau deposition across the overweight/obese and lean groups. These will be measured through the results of the blood tests, MRI scan & data from the PET scans.

CONTACTS AND LOCATIONS:
Overall Officials: Cyrus Raji, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided